CLINICAL TRIAL: NCT02813759
Title: Effect of a Sucralose Preload on Postprandial Metabolic Parameters and Satiety in Subjects With Type 2 Diabetes Mellitus Under Intensive Insulin Therapy - Controlled Clinical Trial
Brief Title: Sucralose in Subjects With Diabetes Mellitus Insulin Requesting
Acronym: SDMIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Claudia Vega Soto, Nutritionist, Universidad de Valparaiso
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17/2015
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GLYCEMIA; SATIETY; C PEPTIDE; PRELOAD; INSULIN
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — trichlorosucrose; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucralose (Experimental): 14 mg sucralose (Zero K sucralose powder, IANSA®) an 200 mL of water
  Interventions: Other: Sucralose
- Water (Placebo Comparator): 200 mL of water
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Sucralose — Subjects drank 200 mL of water with 14 mg sucralose, followed by a standard breakfast.
  Arms: Sucralose
Other: Placebo — Subjects drank 200 mL of water alone (placebo), followed by a standard breakfast.
  Other Names: Water
  Arms: Water

SUMMARY:
To evaluate the acute effect of a preload of sucralose in presence of carbohydrate (HC) available on the glycemic response, postprandial C peptide and satiety in patients with type 2 diabetes mellitus (DM2) in intensive insulin therapy (IIT).

ELIGIBILITY:
Inclusion Criteria:

* Minimum period of six month intensive insulin therapy
* Prescription rapid insulin in the breakfast
* Aged 35 to 70 years
* BMI 25 to 39.9 kg / m2
* HbA1c lower than or equal to 10% (86 mmol / mol)
* Menopausal women under hormone replacement therapy

Exclusion Criteria:

* History of intolerance artificial sweetener sucralose
* Pregnant women
* Puerperal women
* Subjects with neurological disease, endocrine disorder no treatment, kidney disease stage IV or V, cancer, liver disease, chronic obstructive pulmonary disease, HIV
* Subjects with history of stroke , acute myocardial infarction and gastrointestinal resection

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Glycemia | up to 120 minutes
  Glycemia (mg/dL) to -15, 30, 60 and 120 minutes, with respect to breakfast intake.
C peptide | up to 60 minutes
  C-peptide at -15 and 60 minutes with respect to breakfast intake
Satiety | up to 120 minutes
  Visual Analog Scale (VAS) was applied immediate and tardy postprandial (two hours after eating breakfast).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lohner S, Kuellenberg de Gaudry D, Toews I, Ferenci T, Meerpohl JJ. Non-nutritive sweeteners for diabetes mellitus. Cochrane Database Syst Rev. 2020 May 25;5(5):CD012885. doi: 10.1002/14651858.CD012885.pub2. PMID 32449201